CLINICAL TRIAL: NCT06379672
Title: An Investigation of the Efficacy of Resonance Breathing Training in the Rehabilitation of Patients with Long Covid-related Myocardial Injury
Brief Title: Resonance Breathing Training for Long Covid-related Myocardial Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu Sport University (Other)
Responsible Party: Principal Investigator, Ping Yang, Clinical Professor, Chengdu Sport University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023[No.193]
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Long COVID; Myocardial Injury
Keywords: 2D-STE; resonance breathing; Myocardial Injury; Long Covid-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intervention group (Experimental): Subjects were asked to remain in a standing position with their feet shoulder-width apart. The right hand was placed on the chest and the left hand on the abdomen. Inhale to make the abdomen bulge and exhale to make the abdomen sink (inhale through the nose and exhale through the mouth). This was done 2 times a day, once in the morning and once in the afternoon. Complete 3 sets of 8 breaths each. Each breath lasts 10 seconds (4 seconds inhaling and 6 seconds exhaling).
  Interventions: Other: Resonance breathing

INTERVENTIONS:
Other: Resonance breathing — Resonant breathing was used on the subjects, using nasal inhalation and oral exhalation, for a total of 12 weeks.

SUMMARY:
An investigation of the efficacy of resonance breathing training in the rehabilitation of patients with Long covid-related myocardial injury

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60 years;
2. According to the WHO definition: one or more systemic involvement present 3 months after the diagnosis of a new crown infection, and at least 2 of these months cannot be explained by other diseases
3. 2D-STE suggestive of GLSAVG: -17% ≤ men ≤ -10%, -18% ≤ women ≤ -10%;
4. Consent for enrollment based on the degree of myocardial injury, as diagnosed by a clinician;
5. Signing the informed consent form with the consent of the patient or his/her family members

Exclusion Criteria:

* (1) Previous history of coronary atherosclerotic heart disease and heart failure; (2) Combination of severe arrhythmia or cardiogenic shock; (3) Combination of severe hypertension, hypertrophic cardiomyopathy, valvular disease of moderate or higher grade, acute myocarditis or pericarditis; (4) Combination of any disease that severely affects limb movement, such as musculoskeletal system disease or severe hepatic or renal insufficiency; (5) Combination of progressive malignant tumors, infectious diseases, bleeding disorders, autoimmune diseases, etc; Those who have serious mental illness and are unable to cooperate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-25 (Estimated); Primary Completion 2024-09-25 (Estimated); Study Completion 2024-10-05 (Estimated)

PRIMARY OUTCOMES:
New YorkHeart Association (NYHA) | 12weeks
  The scale is divided into four levels
  Grade 1 is unrestricted activity. Daily physical activity does not cause significant shortness of breath, fatigue or palpitations Grade 2 is a mild limitation of activity. Asymptomatic at rest, daily activities may cause significant shortness of breath, fatigue or palpitations Grade 3 is marked limitation of activity. May be asymptomatic at rest, but may cause significant shortness of breath, fatigue, or palpitations with less than daily activity.
  Grade 4 is symptomatic at rest, with discomfort associated with any physical activity. Class IVa for those who can move around indoors or at the bedside without intravenous drug administration; Class IVb for those who cannot get out of bed and require intravenous drug administration.
left ventricle global longitudinal strain, LVGLS | 12weeks
  The magnitude of overall longitudinal myocardial strain in the left ventricle on two-dimensional speckle tracking echocardiograms as an average of the peak longitudinal strain in all myocardial segments. The normal range is (-25% to -17%) in men and (-25% to -18%) in women.

SECONDARY OUTCOMES:
hypertension | 12weeks
  Blood pressure included both systolic and diastolic blood pressure and was observed before and after the intervention for any reduction in blood pressure.
Average heart rate | 12weeks
  One-minute average heart rate (at rest).